CLINICAL TRIAL: NCT01537523
Title: To Investigate the Effect of Early Community-care Program on Physical and Depressive Aspects for Discharged Hospital Patient Suffered From Hip Fracture.
Brief Title: To Investigate the Effect of Early Community-care Program on Fracture Hip Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hong Kong Healthcare Volunteer Organization (Other)
Responsible Party: Principal Investigator, MR L, Chief Executive Officer, Hong Kong Healthcare Volunteer Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RCT-001
Record Dates: First submitted 2012-02-08; First posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Fracture
Keywords: physical; psychological; fracture hip
MeSH Terms: conditions — Fractures, Bone; Hip Fractures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- community-care program (Experimental): receive intervention for 12 weeks
  Interventions: Procedure: community-care program
- control (No Intervention)

INTERVENTIONS:
Procedure: community-care program — community nurse care, physiotherapy
  Arms: community-care program

SUMMARY:
The early community-care program is well-known rehabiliation for the fracture hip patient. For the discharged fracture hip patient from hospital, it is worth to investigate the effect of early mobilization program to improve their physical and psychological aspects.

DETAILED DESCRIPTION:
60 fractured hip patient will randomized allocated into intervention group and control group.

The community-care include nursing care, physiotherapy and home modification according to the condition of the patient.

The intervention will received community-care program for 12 weeks. Two sessions per week and total 24 sessions.

The control group will receive the traditional medication. The outcome measure include elderly mobility scale and happiness scale. The measurement will take at initial and completion of the program.

SPSS will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* fracture hip patients discharged from queen mary hospital

Exclusion Criteria:

* cognitive impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Elderly Mobility Scale | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: HO HO, MSc, Study Director — Volunteer department